CLINICAL TRIAL: NCT00711776
Title: Bioequivalence Study of Aciclovir 5% Cream - Bioequivalence Study of Aciclovir Cream Between Current and New Formulation in Japanese Healthy Volunteers -
Brief Title: Bioequivalence Study of Aciclovir 5% Cream in Japanese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZVC111449
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Herpes Labialis
Keywords: Aciclovir cream 5%; Volunteer; Japanese; Male; Bioequivalence
MeSH Terms: conditions — Herpes Labialis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Subjects receiving new formulation in blank test group (Experimental): Eligible subjects will receive acyclovir cream 5 % following single topical application.
  Interventions: Drug: New formulation
- Subjects receiving current formulation in blank test group (Active Comparator): Eligible subjects will receive acyclovir cream 5 % following single topical application.
  Interventions: Drug: Current formulation
- Subjects receiving new formulation in pre-test group (Experimental): Eligible subjects will receive acyclovir cream 5 % following single topical application.
  Interventions: Drug: New formulation
- Subjects receiving current formulation in pre-test group (Active Comparator): Eligible subjects will receive acyclovir cream 5 % following single topical application.
  Interventions: Drug: Current formulation
- Subjects receiving new formulation in main-test group (Experimental): Eligible subjects will receive acyclovir cream 5 % following single topical application.
  Interventions: Drug: New formulation
- Subjects receiving current formulation in main-test group (Active Comparator): Eligible subjects will receive acyclovir cream 5 % following single topical application.
  Interventions: Drug: Current formulation

INTERVENTIONS:
Drug: New formulation — New formulation of Aciclovir Cream 5% scheduled to be substituted to Current formulation in Japan
  Arms: Subjects receiving new formulation in blank test group; Subjects receiving new formulation in main-test group; Subjects receiving new formulation in pre-test group
Drug: Current formulation — Current formulation of Aciclovir Cream 5% in Japan
  Arms: Subjects receiving current formulation in blank test group; Subjects receiving current formulation in main-test group; Subjects receiving current formulation in pre-test group

SUMMARY:
This study is designed to show bioequivalence between Current and New formulation of Aciclovir cream 5% in keratin layer of the epidermis in Japanese Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese adult males between 20 and 55 years of age, inclusive.

Healthy subjects are defined as individuals who are free from clinically significant disease as determined by their medical history, physical examination, clinical laboratory examinations, vital sign, 12-lead ECG, immunology tests and urinary drug screen test.

* Bodyweight >50 kg and body mass index (BMI) between 18.5 and 28.0 at screening.
* Subjects must be capable of providing written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Baseline QTc interval <450 msec.
* Non-smoker or ex-smoker having ceased smoking for at least 6 months.
* Clinical laboratory examination (AST, ALT, ALP and GGT) at screening are within the normal range.
* The subject is able to attend all visits and complete the study.

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening physical examination, vital sign measurement, 12-lead ECG recording and/or clinical laboratory examination that is deemed by the principal investigator and/or medical monitor to make the subject ineligible for inclusion because of a safety concern.
* History of regular alcohol consumption exceeding, on average, 14 drinks/week (1 drink = 5 ounces (150 mL) of wine or 350 mL of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits) within 6 months of screening.
* Positive for urine drug at screening.
* Positive for syphilis, HIV antibody, Hepatitis B surface antigen, Hepatitis C antibody or HTLV-1 antibody at screening.
* Donation of blood in excess of 400mL within 4 months or 200mL within 1 months prior to at screening.
* History of drug abuse, or current conditions of drug abuse or alcoholism.
* Participation in a clinical study or post-marketing study with an investigational or a non-investigational product or device within 4 months of preceding the first application of study medication.
* Participation in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational or a non-investigational product or device.
* History of asthma, anaphylaxis or anaphylactoid reactions, severe allergic responses.
* The subject has an allergy for any drug or idiosyncrasy. This excludes a pollen allergy without current symptoms.
* At the part obtaining keratinized layer, having exanthem, pigment abnormality, the skin symptoms such as wounds and/or an excessive sunburn.
* History of clinically significant itching, erythema and/or rash by any paster.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-04-10 (Actual); Primary Completion 2008-08-17 (Actual); Study Completion 2008-08-17 (Actual)

PRIMARY OUTCOMES:
Bioequivalence of Aciclovir amount in keratin layer of the epidermis between Current and New formulation of Aciclovir cream | One day

SECONDARY OUTCOMES:
To investigate the safety and tolerability of New and Current formulation of Aciclovir Cream 5% following single topical application in healthy Japanese male subjects | One day

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Results for study ZVC111449 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/ZVC111449?search=study&study_ids=ZVC111449#rs